CLINICAL TRIAL: NCT03775980
Title: CIRSE Emprint Microwave Ablation Registry
Acronym: CIEMAR
Status: Completed | Type: Observational
Sponsor: Cardiovascular and Interventional Radiological Society of Europe (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: CIEMAR
Record Dates: First submitted 2018-12-11; First posted 2018-12-14 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Neoplasms Malignant; Neoplasm Metastasis
MeSH Terms: conditions — Colonic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Emprint Microwave Ablation System — Microwave Ablation of colorectal liver metastases

SUMMARY:
Observation of the clinical use of the Emprint Microwave Ablation System for the ablation of Liver Metastases of Colorectal Adenocarcinoma.

DETAILED DESCRIPTION:
The CIRSE Emprint Microwave Ablation Registry (CIEMAR) is collecting real-life data on the microwave ablation (MWA) of colorectal liver metastatic disease using the Emprint Microwave Ablation System (full study duration) or Emprint HP Microwave Ablation System (from 2021 onwards).

CIEMAR is a prospective, single-arm, multi-centre observational (non-interventional) study with the objective to observe the "real-life" use of MWA in Europe. The study is observing the use of the Emprint or Emprint HP Microwave Ablation System and all patients included in CIEMAR are receiving treatment with this device as their standard care for CRLM.

Primary endpoint: local tumour control in liver at 12 months after MWA on a per lesion basis

Secondary endpoints: Safety; Overall survival; Overall disease-free survival; Hepatic disease-free survival; Time to untreatable progression by thermal ablation; Systemic cancer therapy vacation; Quality of life; Adverse events and toxicity

In order to measure changes in the quality of life of enrolled patients at different moments in time before and after treatment with MWA, CIEMAR is collecting quality of life data using the EORTC QLQ-C30 questionnaire. Filling out the quality-of-life questionnaire is entirely voluntary for the patient. The patient will be offered to fill out the questionnaire in his/her mother tongue.

The site and patient recruitment is complete with 500 patients from 30 sites across 11 European countries. The registry is currently collecting follow-up data (until January 2026).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Proven colorectal liver metastases either histologically proven or diagnosed by imaging in a patient with known colorectal cancer
* Treated with the Emprint or Emprint HP Microwave ablation system
* Patient referred to MWA by a multidisciplinary tumour board
* Signed informed consent form
* Intention to completely treat (ablation, resection, SBRT) all visible disease within 8 weeks
* Maximum number of 9 total liver lesions
* All liver lesions must be local treatment-naive
* Maximum diameter of the largest liver lesion treated with MWA must not exceed 3cm
* Maximum diameter of lesions treated surgically may exceed this limitation
* Maximum number of 5 lung nodules eligible to be treated
* Patients may receive simultaneous liver resection and microwave ablation
* Patients may have received previous systemic therapy
* Patients must not have received surgical resection or thermal ablation for other liver lesions in the last 3 months before inclusion
* Patients treated with a liver-first approach may be included if treatment of the primary tumour is planned
* If applicable: complete response of treated rectal tumour proven by imaging

Exclusion Criteria:

* Life expectancy less than 6 months (palliative treatment)
* Extrahepatic metastases with the exception of a maximum of 5 lung nodules
* Ongoing infection (viral/bacterial)
* Patients receiving simultaneous bowel surgery and microwave ablation
* Patients receiving simultaneous IRE, RFA, SBRT, Cryoablation, HIFU or other local treatment than resection
* Pregnancy
* Patients with liver metastases that cannot be completely and safely treated
* Active cancers other than CRC
* Non-resected primary colon cancer
* Advanced liver disease or evidence of liver insufficiency

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal adenocarcinoma and liver-only or liver-dominant metastatic disease
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2026-01-31 (Actual)

PRIMARY OUTCOMES:
Local Tumor Control | 12 months
  Local Tumor Control at 12 months on a per lesion basis

SECONDARY OUTCOMES:
Number of participants with acute and/or chronic adverse events according to the latest version of CTCAE | 3 years
  Safety and Tolerability will be monitored before, during and after the microwave ablation treatment.
Overall survival | 3 years
  Time from observation until death due to any cause (or censoring)
Overall disease-free-survival | 3 years
  Time from observation until disease progression or death assessed by the investigators
Hepatic disease-free-survival | 3 years
  Time from observation until disease progression in the liver or death assessed by the investigators.
Time to untreatable progression by thermal ablation | 3 years
  Time from the treatment to the point when liver malignancies can no longer be treated by thermal ablation.
Systemic cancer therapy vacation | 3 years
  Time that participants can be removed from systemic cancer therapies following the microwave ablation treatment.
Treatment specific quality of life | 1 year
  Treatment specific quality of life will be assessed using the EORTC-QLQ-C30 questionnaire which includes 28 questions on a scale of 1 to 4 where 1 indicates lower impact of the disease on the patient's quality of life and 4 represents a high impact. Additionally 2 questions using a scale form 1 to 7 are used to generally assess the patient's quality of life where 1 represents poor quality of life and 7 represents an excellent quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Phillippe L. Pereira, PhD, Study Chair — Radiology, Minimally Invasive Therapies and Nuclear Medicine at SLK Clinics Heilbronn GmbH, Germany
Locations (38):
- University Hospital Centre Sisters of Mercy, Zagreb, Croatia
- Aarhus University Hospital, Aarhus, Denmark
- France (3):
  - University Hospital of Nimes, Nîmes
  - CHU de Reims, Reims
  - Les Hôpitaux Universitaires de Strasbourg, Strasbourg
- Germany (12):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Vivantes Klinikum Neukölln, Berlin
  - DRK Kliniken Berlin Westend, Berlin
  - Städtisches Klinikum Braunschweig, Braunschweig
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Krankenhaus Nordwest, Frankfurt
  - Universitätsklinikum Frankfurt, Frankfurt
  - Medizinische Hochschule Hannover, Hanover
  - SLK Kliniken Heilbronn, Heilbronn
  - Krankenhaus Barmherzige Brüder München, Munich
  - Universitätsklinikum Regensburg, Regensburg
  - Tübingen University Hospital, Tübingen
- Attikon University Athens, Athens, Greece
- Italy (7):
  - Fondazione Poliambulanza Brescia, Brescia
  - IRCCS San Giuseppe Multimedica, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - European Institute of Oncology, Milan
  - Ospedaliero Universitaria San Luigi Gonzaga di Orbassano, Orbassano
  - Ospedale Santissima Annunziata, Taranto
  - Città della Salute e della scienza Torino, Torino
- Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania
- Netherlands (3):
  - Amsterdam University Medical Center, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - Leids Universitair Medisch Centrum, Leiden
- City General Hospital 8th September, Skopje, North Macedonia
- Oslo University Hospital, Oslo, Norway
- Portugal (2):
  - Centro Hospitalar Universitário de Lisboa Central, Lisbon
  - IPO Porto, Porto
- Spain (3):
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Turkey (Türkiye) (2):
  - Cukurova University Medical School, Adana
  - Hacettepe University Hospital, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pereira PL, Bale R, Fretland AA, Goldberg SN, Helmberger T, Meijerink MR, Orsi F, Stattner S, Vogl T, Kafkoula A, de Jong N, Zeka B, de Baere T. Local Tumour Control Following Microwave Ablation: Protocol for the Prospective Observational CIEMAR Study. Cardiovasc Intervent Radiol. 2024 Jan;47(1):121-129. doi: 10.1007/s00270-023-03573-0. Epub 2023 Oct 26. PMID 37884801